CLINICAL TRIAL: NCT01154907
Title: Prevention of HIV and Improved Diagnosis of Adolescent Genital Disease in Bilharzia Endemic KwaZulu-Natal, South Africa
Brief Title: Prevention of Female Genital Schistosomiasis (FGS) in Rural High-endemic South Africa
Acronym: VIBE-FGS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Oslo University Hospital (Other)
Collaborators: University of KwaZulu (Other); University of Agder (Other); Sorlandet Hospital HF (Other Government); University of Copenhagen (Other); Leiden University Medical Center (Other); Universiteit Antwerpen (Other)
Responsible Party: Principal Investigator, Eyrun Floerecke Kjetland, MD, Oslo University Hospital
Other Study IDs: VIBE-FGS
Record Dates: First submitted 2010-06-30; First posted 2010-07-01 (Estimated); Last update posted 2017-09-19 (Actual); Status verified 2017-09

CONDITIONS: Uro-genital Schistosomiasis
Keywords: Uro-genital schistosomiasis; Female; South Africa; Rural; Sexually transmitted diseases
MeSH Terms: conditions — Sexually Transmitted Diseases | interventions — Praziquantel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine, stool, blood, in the adults also vaginal lavage and Pap smears
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Girls ages 10-12: In 18 rural schools in Ugu District, South Africa. Undergoing mass-treatment provided by the Department of Health.
  Praziquantel was administered at 40mg/kg in annual mass-treatment
  Interventions: Drug: Praziquantel
- Young adult women: In rural schools in three districts, South Africa. Undergoing mass-treatment provided by the Departments of Health.
  Praziquantel was administered at 40mg/kg in annual mass-treatment
  Interventions: Drug: Praziquantel

INTERVENTIONS:
Drug: Praziquantel — One day, 40mg/kg standard mass Praziquantel as recommended by WHO and local authorities
  Other Names: Biltricide

SUMMARY:
Schistosomiasis is a poverty-related water-transmitted parasitic disease affecting more that 200 million people world wide. Infection with Schistosoma haematobium may cause Female Genital Schistosomiasis (FGS) with pathological lesions in the female genital tract, especially the cervix. Findings indicate that FGS is a hitherto under-diagnosed illness of young women in endemic poor tropical countries, deserving further attention. A cross-sectional study from Zimbabwe indicated that the pathologic genital lesions were unchanged two years after praziquantel treatment in adult women whereas in those who had been treated with praziquantel in childhood the prevalence of genital lesions was significantly lower. Furthermore, a higher prevalence of HIV was detected in women with FGS compared to those without. The proposed project aims at achieving a better understanding of how annual distribution of praziquantel to pre- and post-pubertal schoolgirls may prevent FGS. This information can be of use in current schistosomiasis control programs in the near term resulting in improved strategies for treatment. Preventing or reducing the risk of FGS and genital lesions will lead to improved reproductive health among in women living in schistosomiasis endemic areas.

Project Goal: Contribute to a reduction of the global burden of female genital schistosomiasis (FGS) through improved knowledge about the prevention of gynecological lesions and through improved diagnosis of FGS.

DETAILED DESCRIPTION:
Provide a more extensive description, if desired. Avoid duplication of information to be recorded elsewhere, such as eligibility criteria or outcome measures

ELIGIBILITY:
Inclusion Criteria:

* Females in Schistosoma haematobium endemic areas

Exclusion Criteria:

* Boys
* Pregnancy
* Allergic to praziquantel
* Severe disease

Ages: 10 Years to 23 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: A random sample of school girls in Ugu district, KwaZulu Natal, South Africa
Sampling Method: Probability Sample
Enrollment: 6500 (Estimated)
Dates: Start 2010-04; Primary Completion 2018-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
HIV prevalence after anti-schistosomal treatment in adolescents | 31. December 2021
  HIV prevalence

SECONDARY OUTCOMES:
FGS prevalence and severity after anti-schistosomal treatment in adolescents | 31. December 2021
  Clinical disease
Clinical and laboratory indicators of urogenital schistosomiasis | 31. December 2018
  Polymerase chain reaction (PCR) of vaginal lavage, Cytology, Circulation Anodic Antigen (CAA)

OTHER OUTCOMES:
Pocket Atlas of Female Genital Schistosomiasis | 31. December 2015
  Published by WHO in English, French and Portuguese

CONTACTS AND LOCATIONS:
Overall Officials: Eyrun F Kjetland, MD, PhD, Principal Investigator — Oslo University Hospital, University of KwaZulu-Natal (UKZN); Myra Taylor, PhD, Principal Investigator — UKZN/ Child Development Research Unit (CDRU); Jane Kvalsvig, PhD, Principal Investigator — UKZN/ CDRU; Svein G Gundersen, MD, PhD, Principal Investigator — Agder University Hospital / Sorlandet Hospital
Locations (1):
- University of KwaZulu Natal, Durban, KwaZulu-Natal, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Still collecting and publishing
Supporting Information: Study Protocol, SAP, ICF
Time Frame: December 2021-December 2022
Access Criteria: From endemic country

REFERENCES:
- [Background] Baan M, Galappaththi-Arachchige HN, Gagai S, Aurlund CG, Vennervald BJ, Taylor M, van Lieshout L, Kjetland EF. The Accuracy of Praziquantel Dose Poles for Mass Treatment of Schistosomiasis in School Girls in KwaZulu-Natal, South Africa. PLoS Negl Trop Dis. 2016 May 3;10(5):e0004623. doi: 10.1371/journal.pntd.0004623. eCollection 2016 May. PMID 27139497
- [Background] Bustinduy AL, Friedman JF, Kjetland EF, Ezeamama AE, Kabatereine NB, Stothard JR, King CH. Expanding Praziquantel (PZQ) Access beyond Mass Drug Administration Programs: Paving a Way Forward for a Pediatric PZQ Formulation for Schistosomiasis. PLoS Negl Trop Dis. 2016 Sep 22;10(9):e0004946. doi: 10.1371/journal.pntd.0004946. eCollection 2016 Sep. No abstract available. PMID 27658198
- [Result] Pillay P, van Lieshout L, Taylor M, Sebitloane M, Zulu SG, Kleppa E, Roald B, Kjetland EF. Cervical cytology as a diagnostic tool for female genital schistosomiasis: Correlation to cervical atypia and Schistosoma polymerase chain reaction. Cytojournal. 2016 Apr 20;13:10. doi: 10.4103/1742-6413.180784. eCollection 2016. PMID 27168759
- [Result] Holmen S, Galappaththi-Arachchige HN, Kleppa E, Pillay P, Naicker T, Taylor M, Onsrud M, Kjetland EF, Albregtsen F. Characteristics of Blood Vessels in Female Genital Schistosomiasis: Paving the Way for Objective Diagnostics at the Point of Care. PLoS Negl Trop Dis. 2016 Apr 13;10(4):e0004628. doi: 10.1371/journal.pntd.0004628. eCollection 2016 Apr. PMID 27073857
- [Result] Holmen SD, Kleppa E, Lillebo K, Pillay P, van Lieshout L, Taylor M, Albregtsen F, Vennervald BJ, Onsrud M, Kjetland EF. The first step toward diagnosing female genital schistosomiasis by computer image analysis. Am J Trop Med Hyg. 2015 Jul;93(1):80-86. doi: 10.4269/ajtmh.15-0071. Epub 2015 Apr 27. PMID 25918212
- [Result] Kleppa E, Klinge KF, Galaphaththi-Arachchige HN, Holmen SD, Lillebo K, Onsrud M, Gundersen SG, Taylor M, Ndhlovu P, Kjetland EF. Schistosoma haematobium infection and CD4+ T-cell levels: a cross-sectional study of young South African women. PLoS One. 2015 Mar 13;10(3):e0119326. doi: 10.1371/journal.pone.0119326. eCollection 2015. PMID 25768005
- [Result] Holmen SD, Kjetland EF, Taylor M, Kleppa E, Lillebo K, Gundersen SG, Onsrud M, Albregtsen F. Colourimetric image analysis as a diagnostic tool in female genital schistosomiasis. Med Eng Phys. 2015 Mar;37(3):309-14. doi: 10.1016/j.medengphy.2014.12.007. Epub 2015 Jan 24. PMID 25630808
- [Result] Kildemoes AO, Kjetland EF, Zulu SG, Taylor M, Vennervald BJ. Schistosoma haematobium infection and asymptomatic bacteriuria in young South African females. Acta Trop. 2015 Apr;144:19-23. doi: 10.1016/j.actatropica.2015.01.008. Epub 2015 Jan 24. PMID 25623258
- [Result] Norseth HM, Ndhlovu PD, Kleppa E, Randrianasolo BS, Jourdan PM, Roald B, Holmen SD, Gundersen SG, Bagratee J, Onsrud M, Kjetland EF. The colposcopic atlas of schistosomiasis in the lower female genital tract based on studies in Malawi, Zimbabwe, Madagascar and South Africa. PLoS Negl Trop Dis. 2014 Nov 20;8(11):e3229. doi: 10.1371/journal.pntd.0003229. eCollection 2014. PMID 25412334
- [Result] Kleppa E, Holmen SD, Lillebo K, Kjetland EF, Gundersen SG, Taylor M, Moodley P, Onsrud M. Cervical ectopy: associations with sexually transmitted infections and HIV. A cross-sectional study of high school students in rural South Africa. Sex Transm Infect. 2015 Mar;91(2):124-9. doi: 10.1136/sextrans-2014-051674. Epub 2014 Oct 3. PMID 25281761
- [Result] Kjetland EF, Norseth HM, Taylor M, Lillebo K, Kleppa E, Holmen SD, Andebirhan A, Yohannes TH, Gundersen SG, Vennervald BJ, Bagratee J, Onsrud M, Leutscher PD. Classification of the lesions observed in female genital schistosomiasis. Int J Gynaecol Obstet. 2014 Dec;127(3):227-8. doi: 10.1016/j.ijgo.2014.07.014. Epub 2014 Aug 13. No abstract available. PMID 25179171
- [Result] Kleppa E, Ramsuran V, Zulu S, Karlsen GH, Bere A, Passmore JA, Ndhlovu P, Lillebo K, Holmen SD, Onsrud M, Gundersen SG, Taylor M, Kjetland EF, Ndung'u T. Effect of female genital schistosomiasis and anti-schistosomal treatment on monocytes, CD4+ T-cells and CCR5 expression in the female genital tract. PLoS One. 2014 Jun 4;9(6):e98593. doi: 10.1371/journal.pone.0098593. eCollection 2014. PMID 24896815
- [Result] Pillay P, Taylor M, Zulu SG, Gundersen SG, Verweij JJ, Hoekstra P, Brienen EA, Kleppa E, Kjetland EF, van Lieshout L. Real-time polymerase chain reaction for detection of Schistosoma DNA in small-volume urine samples reflects focal distribution of urogenital Schistosomiasis in primary school girls in KwaZulu Natal, South Africa. Am J Trop Med Hyg. 2014 Mar;90(3):546-52. doi: 10.4269/ajtmh.13-0406. Epub 2014 Jan 27. PMID 24470560
- [Result] Hegertun IE, Sulheim Gundersen KM, Kleppa E, Zulu SG, Gundersen SG, Taylor M, Kvalsvig JD, Kjetland EF. S. haematobium as a common cause of genital morbidity in girls: a cross-sectional study of children in South Africa. PLoS Negl Trop Dis. 2013;7(3):e2104. doi: 10.1371/journal.pntd.0002104. Epub 2013 Mar 21. PMID 23556009
- [Result] Galappaththi-Arachchige HN, Amlie Hegertun IE, Holmen S, Qvigstad E, Kleppa E, Sebitloane M, Ndhlovu PD, Vennervald BJ, Gundersen SG, Taylor M, Kjetland EF. Association of Urogenital Symptoms with History of Water Contact in Young Women in Areas Endemic for S. haematobium. A Cross-Sectional Study in Rural South Africa. Int J Environ Res Public Health. 2016 Nov 14;13(11):1135. doi: 10.3390/ijerph13111135. PMID 27854250
- [Derived] Lothe A, Zulu N, Oyhus AO, Kjetland EF, Taylor M. Treating schistosomiasis among South African high school pupils in an endemic area, a qualitative study. BMC Infect Dis. 2018 May 25;18(1):239. doi: 10.1186/s12879-018-3102-0. PMID 29801483
- See also: Project website — http://brightresearch.org
- See also: WHO pocket atlas for Female Genital Schistosomiasis — http://who.int/schistosomiasis/en/